CLINICAL TRIAL: NCT05386589
Title: An Open-Label, Single-Dose Clinical Study to Evaluate the Pharmacokinetics of Molnupiravir (MK-4482) in Participants With Moderate Hepatic Impairment
Brief Title: A Study to Evaluate Molnupiravir (MK-4482) in Participants With Moderate Hepatic Impairment (MK-4482-016)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4482-016; MK-4482-016 (Other: MSD)
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Results first posted 2024-05-09 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — molnupiravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment received a single oral dose of molnupiravir 800 mg on Day 1.
  Interventions: Drug: Molnupiravir
- Healthy-Matched Control Group (Experimental): Healthy matched participants received a single oral dose of molnupiravir 800 mg on Day 1.
  Interventions: Drug: Molnupiravir

INTERVENTIONS:
Drug: Molnupiravir — Four 200 mg capsules administered orally as a single dose
  Other Names: MK-4482,; MOV; EIDD-2801

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) of N-hydroxycytidine (NHC) following a single oral dose of molnupiravir in participants 18 to 75 years (inclusive) with moderate hepatic impairment and healthy matched controls.

ELIGIBILITY:
The key inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has a BMI ≥18.5 and ≤35 kg/m2
* Diagnosis of chronic (>6 months) stable Hepatic Impairment (HI) with features of cirrhosis due to any etiology (Moderate HI arm only)
* Has a score on the Child-Pugh scale ranging from 7 to 9 (Moderate HI arm only)
* In good health (except for Moderate HI)

Exclusion Criteria:

* Anticipated survival of <3 months (Moderate HI arm only)
* Received antiviral and/or immune modulating therapy (Moderate HI only) for Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) within 90 days prior to study start
* History of clinically significant abnormalities or diseases (Healthy matched arm only).
* History of cancer
* Major surgery and/or donated or lost 1 unit of blood
* Taking medications to treat chronic medical conditions and has not been on a stable regimen for at least 1 month (Moderate HI arm only) and/or is unable to withhold the use of the medication(s) within 4 hours prior to and 8 hours after administration of the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2023-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (3):
- United States (3):
  - Research Centers of America ( Hollywood ) ( Site 0002), Hollywood, Florida
  - Clinical Pharmacology of Miami ( Site 0003), Miami, Florida
  - Thomas Jefferson University - Pharmacology and Experimental Therapeutics ( Site 0001), Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Duncan KE, Carstens RP, Butterfield KL, Jin Y, Inbody LR, Schaeffer AK, Matthews CZ, Zhao T, Patel S, Maas BM, Cheng MH, Stoch SA. Assessment of pharmacokinetics and tolerability following single-dose administration of molnupiravir in participants with hepatic or renal impairment. Clin Transl Sci. 2024 Dec;17(12):e70073. doi: 10.1111/cts.70073. PMID 39601078
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 3 sites in the United States.
Groups:
- Moderate Hepatic Impairment: Participants with moderate hepatic impairment will receive a single oral 800mg dose of molnupiravir.
- Healthy-Matched Control Group: Healthy matched participants will receive a single oral 800mg dose of molnupiravir.
Period: Overall Study
Arm/Group | Moderate Hepatic Impairment | Healthy-Matched Control Group
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Hepatic Impairment | Healthy-Matched Control Group | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (10.2) | 54.6 (2.9) | 54.3 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-∞) of Plasma N-Hydroxycitidine (NHC)
Description: The plasma AUC0-∞ of NHC is reported.
Time Frame: Day 1: Predose and 0.5, 1.5, 2, 4, 6, 8, 12, 24, 48, and 72 hours postdose
Population: All participants are included.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/mL
Arm/Group | Moderate Hepatic Impairment | Healthy-Matched Control Group
Number analyzed (Participants) | 7 | 7
hr*ng/mL | 8930 [6560 to 12100] | 10900 [8510 to 14000]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of NHC
Description: The plasma Cmax of NHC is reported.
Time Frame: Day 1: Predose and 0.5, 1.5, 2, 4, 6, 8, 12, 24, 48, and 72 hours postdose
Population: All participants are included.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Moderate Hepatic Impairment | Healthy-Matched Control Group
Number analyzed (Participants) | 7 | 7
ng/mL | 3660 [2730 to 4900] | 3790 [3260 to 4420]

3. Secondary Outcome: Number of Participants Experiencing ≥1 Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to ~ 14 days
Population: All participants are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hepatic Impairment | Healthy-Matched Control Group
Number analyzed (Participants) | 7 | 7
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to ~14 days
Description: All participants are included.
Arm/Group | Moderate Hepatic Impairment | Healthy-Matched Control Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate Hepatic Impairment (N=7) | Healthy-Matched Control Group (N=7)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT05386589/Prot_SAP_000.pdf